CLINICAL TRIAL: NCT05251051
Title: Project INITIATE: Developing Community Collaborations to Improve Developmental Outcomes Through Prompt and Equitable Transition to Community Therapy Services in High-risk Newborn Infants
Brief Title: Project Initiate: Transition to Community Therapy Services After NICU Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Raye Ann deRegnier, Professor of Pediatrics, Northwestern University Feinberg School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-4541
Record Dates: First submitted 2022-01-28; First posted 2022-02-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Motor Delay
MeSH Terms: conditions — Psychomotor Disorders

STUDY DESIGN:
Intervention Model Description: Infants will be assigned to an intervention or control group based on the city of residence at discharge (Chicago or not-Chicago)
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by blinded neuromotor examiners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): At NICU discharge, infants will be referred to Illinois Early Intervention. A coordinator (the navigator) will assist families in engaging with Early Intervention and completing all enrollment requirements.
  At NICU discharge, infants will be provided with standard home pediatric therapy services weekly for up to 14 weeks. These will be initiated within 2 weeks of discharge.
  Interventions: Behavioral: pediatric physical therapy; Other: Care Coordination
- Control Group (Other): At NICU discharge, infants will be referred to Illinois Early Intervention. A coordinator (the navigator) will assist families in engaging with Early Intervention and completing all enrollment requirements. If transitional services were recommended by the NICU providers, the navigator will help families identify these services and obtain the necessary referrals.
  Interventions: Other: Care Coordination

INTERVENTIONS:
Behavioral: pediatric physical therapy — Pediatric physical therapists will provide weekly home therapy using standard of care/best evidence procedures
  Arms: Intervention Group
Other: Care Coordination — A navigator will be assigned who will assist families in obtaining Early Intervention services and other therapy services if needed
  Other Names: Navigation

SUMMARY:
Project Initiate is a pilot study of early neuromotor outcomes in high risk newborn infants who are referred to Early Intervention services after NICU discharge. The investigators hypothesize that infants with Medicaid insurance who have prompt access to weekly post-discharge therapy services will have better early neuromotor function at 3 months corrected age and better parent satisfaction than infants who receive only care coordination to help with Early Intervention enrollment and locating outpatient transitional services as indicated.

DETAILED DESCRIPTION:
Infants hospitalized in an neonatal intensive care unit with high risk illnesses typically receive physical therapy during the hospital stay to improve neuromotor function and promote optimal development. At discharge, infants residing in Illinois with high risk conditions are eligible for therapy services in the home through Illinois Early Intervention. The initiation of these services is typically delayed for several months or more after discharge and families with private insurance will often obtain transitional services. For children with Medicaid insurance, initiation of services is typically delayed or never occurs and there is concern that gaps in services may worsen outcomes and cause stress to parents.

The investigators hypothesize that infants with Medicaid insurance who have prompt access to weekly post-discharge therapy services will have better early neuromotor function at 3 months corrected age and better parent satisfaction than infants who receive only care coordination to help with Early Intervention enrollment and locating outpatient transitional services as indicated.

The aims of Project Initiate are:

Specific Aim 1: To pilot a NICU to home service delivery model for infants at high-risk for neuromotor complications with Medicaid Insurance.

Specific Aim 2: To test the feasibility of at NICU to home service delivery model for infants at high-risk for neuromotor complications.

Specific Aim 3: To compare motor and parental quality of life outcomes at 3-4 months corrected age in study participants and those who received standard discharge services.

Families of infants with high risk medical conditions qualifying for Early Intervention services will be recruited at NICU discharge and assigned to the intervention or control group based on the parents' city of residence (based on the availability of home therapists by location).

For the intervention group, therapy will be provided weekly within two weeks of discharge. Infants will be enrolled in Early Intervention, infants will receive care coordination to assist in engagement with the Early Intervention program and home services will be provided through the study until the Early intervention services are fully engaged or for 14 weeks, whichever comes first.

For the control group, infants will be enrolled in Early Intervention and infants will receive care coordination to assist in engagement with the Early Intervention program. If transitional services are recommended at discharge, the therapy care coordinator will assist families with these referrals until Early intervention is fully engaged r for 14 weeks, whichever comes first.

At discharge, neuromotor outcomes will be assessed. At 3 months corrected age, all infants will be evaluated in the Early Childhood clinic and their neuromotor outcome will be assessed. Parents will also complete quality of life surveys at discharge and at 3 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

At-risk for developmental impairments (enrolled in Early Childhood Clinic and are automatically eligible for Illinois Early Intervention services)

Less that 45 weeks post-menstrual age (PMA) at discharge

English-speaking

Able to be identified and enrolled before discharge from the NICU

Exclusion Criteria:

Children in DCFS custody or children of parents who decline therapy services through the State of Illinois Early Intervention Program.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Test of Infant Motor Performance Score (TIMP) | 2-3 months (discharge to first developmental clinic visit)
  The TIMP is a motor evaluation conducted by a physical therapist. The test is scored and the scores are converted to standard deviations based on the child's age. Changes in the infant's TIMP standard deviation score from discharge to 3 months of age, corrected for prematurity, assessed by an physical therapist blinded to the intervention group.
Time to initiation of Early Intervention therapy services | Discharge to EI initiation (1-6 months)
  The time from discharge to the first Early Intervention home therapy service will be assessed
Parent quality of life questionnaire assessed using the Peds QL Family Impact Module | 2-3 months
  Parent quality of life will be assessed at the beginning and end of the study. This test asks parents to rate their quality of life in 6 categories. Each item is scored on a Likert Scale from 0-4 and then reverse transformed to a score from 0-100. The investigators will use an overall score averaged from the 6 categories as an outcome, as well as scores for the individual categories. Higher scores indicated better parent reported quality of life.

SECONDARY OUTCOMES:
General movements assessment- | At 3 months corrected age
  Motor optimality scores will be obtained from observation of standard videos and rated by blinded trained observers. Motor optimality scores can range from 5-28 with higher scores indicating better motor optimality.
Hammersmith Infant Neurologic examination | At 3 months corrected age
  A neurologic examination performed by blinded observers who have been trained (physical therapists or physicians). Each item (n=26) is scored from 0-3 points. Higher scores indicate better neurologic function with a maximum score of 78.

CONTACTS AND LOCATIONS:
Overall Officials: Raye-Ann deRegnier, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - University of Illinois at Chicago, Chicago, Illinois
  - Lurie Children's Hospital, Chicago, Illinois
  - Prentice Women's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No